CLINICAL TRIAL: NCT02841501
Title: Genetic Susceptibility Factors Involved in Candidemia: Case-control Study.
Brief Title: Genetic Susceptibility Factors for Candidemia.
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Seventh Framework Programme (Other); University of Lausanne Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: 2011_63; 2012-A01344-39 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-07-20; First posted 2016-07-22 (Estimated); Last update posted 2021-03-26 (Actual); Status verified 2020-08

CONDITIONS: Invasive Candidiasis; Candidemia; Genetic Predisposition to Disease
Keywords: Gene Expression Profiling; Genome-Wide Association Study; Polymorphism, Single Nucleotide; Drug Resistance, Fungal
MeSH Terms: conditions — Candidiasis, Invasive; Candidemia; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 20 mL of blood samples are collected at inclusion. 10 mL on EDTA tubes for the genetic analysis, and 1 mL on dry tube for biomarkers development.
  Paxgen tubes will be collected in a sample of patients for a transcriptomic study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Candidemia patients: These patients are included in the study after the reception of a positive blood culture for Candida sp.
  Interventions: Genetic: Analysis of genetic polymorphisms
- Control patients: These patients are matched on case patients on the following criteria:
  * Age+/-5 years
  * length of hospitalisation
  * type of ward
  * type of surgery for surgical patients
  * IGS2 for intensive care patients
  Interventions: Genetic: Analysis of genetic polymorphisms

INTERVENTIONS:
Genetic: Analysis of genetic polymorphisms — An analysis of the SNPs (single nucleotide polymorphism) of 25 candidate genes will be performed. This analysis will be completed by a genome wide association study.

SUMMARY:
This is a prospective case-control physiopathological study, which main objective is to determine the genetic host factors predisposing to candidemia. Secondary objectives are to develop new diagnosis tools using the biological collection, to describe and update epidemiology, to analyse the influence of genetic polymorphisms on prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years.
* Informed consent.
* Positive blood culture with isolation of Candida sp.

Exclusion Criteria:

* No informed consent.
* Patient younger than 18.
* No insurance coverage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients exhibiting a positive blood culture with isolation of Candida sp.
Sampling Method: Non-Probability Sample
Enrollment: 453 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Frequency of the polymorphisms between the groups | In the 48-72 hours following the positive blood culture

CONTACTS AND LOCATIONS:
Overall Officials: Julien Poissy, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Salengro, Intensive care departement, CHRU, Lille, France

IPD SHARING:
Plan to Share IPD: No